CLINICAL TRIAL: NCT02865720
Title: A Phase 3, Open-label, Single-period Study to Evaluate the Safety and Treatment Effect of Intravenous Administration of C1 Inhibitor (Human) for the Prevention of Angioedema Attacks and Treatment of Breakthrough Attacks in Japanese Subjects With Hereditary Angioedema (HAE)
Brief Title: Study of C1 Inhibitor (Human) for the Prevention of Angioedema Attacks and Treatment of Breakthrough Attacks in Japanese Subjects With Hereditary Angioedema (HAE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP616-209; 0624-209 (Other: Shire)
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — SERPING1 protein, human

ARMS (2):
- Subjects 2 to 5 years of age (Experimental): 500 U of CINRYZE will be administered by IV infusion twice weekly for 12 weeks
  Interventions: Drug: CINRYZE 500 U
- Subjects 6 years of age and older (Experimental): 1000 U of CINRYZE will be administered by IV infusion twice weekly for 12 weeks.
  Interventions: Drug: CINRYZE 1000 U

INTERVENTIONS:
Drug: CINRYZE 500 U — IV infusion administered twice weekly
  Arms: Subjects 2 to 5 years of age
Drug: CINRYZE 1000 U — IV infusion administered twice weekly
  Arms: Subjects 6 years of age and older

SUMMARY:
The purpose of this study is to determine if an investigational treatment is safe and well tolerated when administered by intravenous (IV) infusion in Japanese subjects with HAE.

ELIGIBILITY:
Inclusion Criteria:

1. Be of Japanese descent, defined as born in Japan and having Japanese parents and Japanese maternal and paternal grandparents.
2. Be ≥2 years of age.
3. Meet the following minimum body weight criteria:

   * Subjects 2 to 5 years of age must weigh at least 12.5 kg; and
   * Subjects 6 years of age and above must weigh at least 25 kg.
4. Have a confirmed diagnosis of Type I or Type II HAE. NOTE: Diagnosis may be based on historical data including family history, clinical symptoms (characteristic attacks), or documentation of low level of C1 INH protein and/or C1 INH activity.
5. Have a history of at least one angioedema attack per month (on average) during the 3 consecutive months immediately before enrollment.
6. Agree to adhere to the protocol-defined schedule of assessments and procedures.
7. Agree to avoid his/her known angioedema attack triggers during the study to the best of his/her ability.
8. If a female of reproductive age, be postmenopausal (≥12 months following cessation of menstruation), surgically sterile, or following an acceptable method of birth control (and agree to continue its use through 1 month after the last dose of study drug):

   * Non-hormonal methods (eg, abstinence, barrier control) for at least 1 complete menstrual cycle before the Screening Visit.
   * Stable doses of estrogen and/or progestin containing products for at least 2 months before the Screening Visit.
9. If a male of reproductive age, be surgically sterile or agree to follow an acceptable method of birth control (eg, abstinence, barrier control) from the Screening Visit through 2 months after the last dose of study drug.
10. If an adult, be informed of the nature of the study and provide written informed consent before any study-specific procedures are performed.

OR If a child or minor (<20 years of age), have a parent/legal guardian who is informed of the nature of the study provide written informed consent (ie, permission) for the child to participate in the study before any study-specific procedures are performed. Assent will be obtained from children ≥14 years of age.

Exclusion Criteria:

1. Have a history of hypercoagulability (abnormal blood clotting).
2. Have a diagnosis of acquired angioedema or be known to have C1 INH antibodies.
3. Have a history of allergic reaction to C1 INH products, including CINRYZE (or any of the components of CINRYZE) or other blood products.
4. Have received C1 INH therapy or any blood products within 3 days before the first dose of study drug.
5. Have had signs or symptoms of an angioedema attack within 2 days before the first dose of study drug.
6. Have any change (start, stop, or change in dose) in androgen therapy (eg, danazol, oxandrolone, stanozolol, testosterone), tranexamic acid, epsilon-aminocaproic acid (EACA), or other antifibrinolytics within 14 days before the first dose of study drug.
7. If female, have started taking or changed the dose of any hormonal contraceptive regimen or hormone replacement therapy (eg, estrogen/progestin containing products) within 2 months before the first dose of study drug.
8. Be pregnant or breastfeeding.
9. Have received an investigational drug other than those required for prevention or treatment of angioedema attacks within 30 days before the first dose of study drug.
10. Have, as determined by the Investigator and/or the Sponsor's Medical Monitor, any surgical or medical condition that could interfere with the administration of study drug or interpretation of study results.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- Japan (10):
  - Toyohashi Municipal Hospital, Toyohashi, Aiti
  - Asahi General Hospital, Asahi, Chiba
  - Gunma University Hospital, Maebashi, Gunma
  - Kobe University Hospital, Kobe, Hyōgo
  - Heart Life Hospital, Nakagusuku, Nakagami
  - Naha City Hospital, Naha, Okinawa
  - Shiman University Hospital, Izumo, Shimane
  - Adachi kyosai Hospital, Adachi City, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Tomakomai City Hospital, Tomakomai

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 9 study centers in Japan between 13 Sep 2016 (First participant first visit) and 23 June 2017 (Last participant last visit).
Pre-assignment Details: A total of 8 participants were screened and enrolled. Investigational product administrations were planned according to participants' age; 500 units (U) for participants 2 to 5 years and 1000 U for participants 6 years and older. However, as no participants under the age of 6 years were enrolled, only the higher dose of 1000 U was administered.
Groups:
- CINRYZE 500 U: Participants received 500 U CINRYZE intravenous (IV) injection twice weekly for 12 weeks.
- CINRYZE 1000 U: Participants received 1000 U CINRYZE IV injection twice weekly for 12 weeks.
Period: Overall Study
Arm/Group | CINRYZE 500 U | CINRYZE 1000 U
Started | 0 | 8
Completed | 0 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat safety (ITT-S) set included participants who received any amount of investigational product.
Groups:
- CINRYZE 500 U: Participants received 500 U CINRYZE IV injection twice weekly for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | CINRYZE 500 U | CINRYZE 1000 U | Total
Number analyzed (Participants) | 0 | 8 | 8
Age, Continuous [Mean (Standard Deviation); unit: year] |  | 38.4 (7.27) | 38.4 (7.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 6 | 6
  Male |  | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 8 | 8
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 8 | 8
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 0 | 0
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered an investigational product and that did not necessarily have a causal relationship with the treatment. TEAEs were defined as all AEs that started during the treatment period and up to 7 days after the last dose of investigational product, or AEs that were seen at baseline but worsened in frequency and/or severity during the treatment period and up to 7 days after the last dose of investigational product.
Time Frame: From start of study drug administration up to Week 12
Population: ITT-S set included participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants | 7

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination Reported as Adverse Events (AEs)
Description: Physical examinations included measurement of body weight and height. Clinically significant abnormalities related to physical examination as determined by investigator were recorded and reported as AE.
Time Frame: From start of study drug administration up to Week 12
Population: ITT-S set included participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Vital Signs Reported as Adverse Events (AEs)
Description: Vital sign assessments included systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate. Investigator used both absolute values and change from baseline values to determine if the vital sign was potentially clinically important. Criteria for the potential clinical importance of both absolute and change from baseline values were pre-specified as: SBP (less than [<] 90 millimeter of mercury [mmHg]; greater than or equal to [>=] 140 mmHg), DBP (< 60 mmHg; >=90 mmHg) and pulse (less than or equal to [<=] 50 beats per minute [bpm]; >= 100 bpm. A participant's vital sign had to meet both the absolute and change from baseline criteria to be considered as potentially clinically important.
Time Frame: Baseline up to Week 12
Population: ITT-S set included participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Important (PCI) Clinical Laboratory Assessments Reported as Adverse Events (AEs)
Description: Number of participants with potentially clinically important (PCI) clinical laboratory assessments reported as adverse events were reported.
Time Frame: Baseline up to Week 12
Population: ITT-S set included participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants | 0

5. Primary Outcome: Concentration of C1 Esterase Inhibitor (C1 INH) Antigen (Protein Volume) at Week 1
Description: C1 INH antigen concentration in plasma was determined using an automated nephelometric assay.
Time Frame: Week 1: Pre-dose, 0.5, 1, 2, 6, 24, 48, 72 and 96 hours (h) post-dose
Population: Pharmacokinetic (PK) set included all participants with evaluable PK profiles.
Measure: Mean (Standard Deviation); unit: Gram per liter (g/L)
Groups:
- CINRYZE 1000U: Participants received 1000 U CINRYZE IV injection twice weekly for 12 weeks.
Arm/Group | CINRYZE 1000U
Number analyzed (Participants) | 8
Gram per liter (g/L)
  Pre-dose: number analyzed (Participants) | 7
  Pre-dose | 0.0581 (0.04877)
  0.5 h post-dose: number analyzed (Participants) | 7
  0.5 h post-dose | 0.1463 (0.04210)
  1 h post-dose: number analyzed (Participants) | 5
  1 h post-dose | 0.1426 (0.05795)
  2 h post-dose: number analyzed (Participants) | 7
  2 h post-dose | 0.1436 (0.04524)
  6 h post-dose: number analyzed (Participants) | 6
  6 h post-dose | 0.1413 (0.04376)
  24 h post-dose: number analyzed (Participants) | 7
  24 h post-dose | 0.1147 (0.03825)
  48 h post-dose | 0.0978 (0.04204)
  72 h post-dose: number analyzed (Participants) | 7
  72 h post-dose | 0.0881 (0.04133)
  96 h post-dose: number analyzed (Participants) | 1
  96 h post-dose | 0.0680 (NA) — Standard Deviation is not calculated due to a single participant being evaluable.

6. Primary Outcome: Concentration of C1 Esterase Inhibitor (C1 INH) Antigen (Protein Volume) at Week 12
Description: C1 INH antigen concentration in plasma was determined using an automated nephelometric assay.
Time Frame: Week 12: Pre-dose, 0.5, 1, 2, 6, 24, 48, 72 and 96 h post-dose
Population: PK set included all participants with evaluable PK profiles.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
gram per liter (g/L)
  Pre-dose | 0.0775 (0.04904)
  0.5 h post-dose | 0.1660 (0.04159)
  1 h post-dose: number analyzed (Participants) | 5
  1 h post-dose | 0.1468 (0.03232)
  2 h post-dose | 0.1634 (0.04500)
  6 h post-dose | 0.1573 (0.03978)
  24 h post-dose | 0.1244 (0.04675)
  48 h post-dose | 0.1003 (0.05030)
  72 h post-dose | 0.0836 (0.05169)
  96 h post-dose | 0.0661 (0.05163)

7. Primary Outcome: Concentration of Plasma Complement C4 at Week 1
Description: Concentration of plasma complement C4 was reported.
Time Frame: Week 1: Pre-dose, 0.5, 1, 2, 6, 24, 48, 72 and 96 h post-dose
Population: Pharmacodynamic (PD) set included all participants with evaluable PD profiles.
Measure: Mean (Standard Deviation); unit: Milligram per liter (mg/L)
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Milligram per liter (mg/L)
  Pre-dose | 42.8 (20.42)
  0.5 h post-dose | 37.5 (17.55)
  1 h post-dose: number analyzed (Participants) | 6
  1 h post-dose | 32.7 (18.17)
  2 h post-dose | 43.3 (19.48)
  6 h post-dose | 69.0 (29.70)
  24 h post-dose | 89.0 (33.80)
  48 h post-dose | 82.5 (36.00)
  72 h post-dose | 80.5 (41.34)
  96 h post-dose: number analyzed (Participants) | 1
  96 h post-dose | 67.0 (NA) — Standard Deviation is not calculated due to a single participant being evaluable.

8. Primary Outcome: Concentration of Plasma Complement C4 at Week 12
Description: Concentration of plasma complement C4 was reported.
Time Frame: Week 12: Pre-dose, 0.5, 1, 2, 6, 24, 48, 72 and 96 h post-dose
Population: PD set included all participants with evaluable PD profiles.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
mg/L
  Pre-dose | 77.9 (37.79)
  0.5 h post-dose | 65.0 (37.92)
  1 h post-dose: number analyzed (Participants) | 5
  1 h post-dose | 41.4 (13.79)
  2 h post-dose | 67.5 (40.19)
  6 h post-dose | 91.1 (49.98)
  24 h post-dose | 104 (53.35)
  48 h post-dose | 99.3 (50.65)
  72 h post-dose | 77.9 (47.39)
  96 h post-dose | 63.2 (37.06)

9. Primary Outcome: Concentration of Plasma Complement C1q at Week 1
Description: Concentration of plasma complement C1q was reported.
Time Frame: Baseline (Week 1)
Population: PD set included all participants with evaluable PD profiles.
Measure: Mean (Standard Deviation); unit: International units per milliliter
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
International units per milliliter | 78.50 (36.598)

10. Primary Outcome: Normalized Number of Angioedema Attacks (NNA) Per Month
Description: Angioedema attack was defined as any participant-reported (or caregiver-reported) indication of swelling or pain at any location following a report of no swelling or pain on the previous day (that is, there must have been a full symptom-free calendar day preceding the onset of symptoms for an attack to be considered a new attack). NNA was calculated as the overall number of angioedema attacks recorded during the period divided by the number of days in the period and multiplied by 30.4.Number of attacks was normalized for the number of days participants participated in a given period and expressed as the monthly frequency as compared to the historical data where, NNA was the number of angioedema attacks during 3 months prior to study drug administration. Historical data was obtained from medical or angioedema history electronic case report forms (eCRF).
Time Frame: Baseline up to Week 12
Population: Full analysis set (FAS) included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Angioedema attacks per month
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Angioedema attacks per month
  Historical | 3.375 (2.5225)
  CINRYZE Treatment | 1.826 (1.5031)

11. Primary Outcome: Number of Participants With Angioedema Attacks in Different Anatomic Locations
Description: Anatomic locations where there was a presence of pain or swelling of any level of severity; mild, moderate or severe at any day during the attack were reported. Mild: the attack symptoms were noticeable but were easily tolerated by the participant and did not interfere with the participant's daily activities. Moderate: the attack symptoms interfered with the participant's ability to attend work/school or participate in family life and social/recreational activities and severe: the attack symptoms significantly limited the participant's ability to attend work/school or participate in family life and social/recreational activities. Number of participants with angioedema attacks in different anatomic locations in treatment period was compared to NNA for historical data. Historical data was based on the typical location of angioedema attacks in the 3 months prior to study drug administration. Here, H refers to historical and T refers to treatment.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants
  Abdominal/Gastrointestinal: H | 7
  Abdominal/Gastrointestinal: T | 3
  Cutaneous - Facial: H | 3
  Cutaneous - Facial: T | 2
  Cutaneous - Extremity or Peripheral: H | 6
  Cutaneous - Extremity or Peripheral: T | 6
  Genital/Urinary (Includes scrotum or vulva): H | 2
  Genital/Urinary (Includes scrotum or vulva): T | 4
  Upper Airway (includes laryngeal or pharyngeal): H | 2
  Upper Airway (includes laryngeal or pharyngeal):T | 1

12. Primary Outcome: Average Severity (Intensity) of Angioedema Attacks
Description: All attacks in each therapy period were assigned a value of 1 (mild), 2 (moderate), or 3 (severe). Attack severity was considered the highest value assigned by the participant to any swelling location on any day during the attack. The average severity was derived by dividing the cumulative severity score by the total number of attacks. Average severity was set to 0 if there was no attack in a period. Average severity of angioedema attacks in treatment period compared to the NNA of angioedema attacks for historical data was reported. Historical data was based on the typical severity of angioedema attacks in the 3 months prior to study drug administration. Historical data was obtained from medical or angioedema history electronic case report forms (eCRF).
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Units on a scale
  Historical | 1.875 (0.8345)
  CINRYZE Treatment | 0.970 (0.6441)

13. Primary Outcome: Average Duration of Angioedema Attacks
Description: Average duration of attacks was calculated by dividing the cumulative duration of attacks by the total number of attacks during the treatment period. Historical data was based on the typical severity of angioedema attacks in the 3 months prior to study drug administration. Average duration of angioedema attacks in treatment period was compared to the NNA for historical data. Historical data was obtained from medical or angioedema history eCRF.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Days
  Historical | 2.250 (1.0351)
  CINRYZE Treatment | 1.941 (2.0630)

14. Primary Outcome: Normalized Number of Angioedema Attacks (NNA) Per Month Treated With Rescue Medication
Description: The normalized number of angioedema attacks was calculated as the overall number of angioedema attacks recorded during the period divided by the number of days in the period and multiplied by 30.4. NNA treated with rescue medications were reported for CINRYZE, non-CINRYZE C1-INH or not treated with C1-INH (including attacks treated with any medications other than C1-INH or untreated attacks). CINRYZE was only considered as a rescue medication when treated for breakthrough attack treatment. For historical data, only medications taken prior to the start of drug study drug administration and had an indication of "hereditary angioedema (HAE) management - acute treatment" selected on the prior and concomitant medications and therapy were considered as rescue medications. Historical data was obtained from medical or angioedema history eCRF.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Angioedema attacks per month
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Angioedema attacks per month
  Historical Data | 1.750 (2.2660)
  CINRYZE Treatment | 0.477 (0.8411)

15. Primary Outcome: Number of Participants Achieving Clinical Responder Rate Relative to Historical Data
Description: Number of participants achieving at least 50 percent (%), 70% or 90% reduction in NNA relative to NNA for historical data was reported.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants
  Achieving >= 50% reduction in NNA | 4
  Achieving >= 70% reduction in NNA | 3
  Achieving >= 90% reduction in NNA | 2

16. Primary Outcome: Change From Baseline in Angioedema Quality of Life (AE-QoL) in Treatment Period
Description: Angioedema quality of life (AE-QoL) questionnaire was a self-administered validated angioedema disease-specific quality of life instrument. It consisted of 17 specific questions that were associated with work, physical activity, free time, social relations, and diet. Each of the 17 items had a 5-point response scale ranging from 1 (Never) to 5 (Very Often). The questionnaire was scored according to the developers' guidelines to produce a total score and 4 domain scores (functioning, fatigue/mood, fear/shame, nutrition). Raw domain scores (mean of the item scores within each scale) and the raw total score (mean of all item scores) were rescaled using linear transformations into final percentage scores ranging 0 to 100, based on the maximum possible score, where the higher the score the greater the QoL impairment.
Time Frame: Baseline, Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Score on a scale
  Total Score (Baseline) | 28.3 (12.79)
  Total Score (Change from baseline) | -9.0 (16.72)
  Functioning (Baseline) | 16.4 (11.54)
  Functioning (Change from baseline) | -2.3 (22.39)
  Fatigue/Mood (Baseline) | 18.8 (19.59)
  Fatigue/Mood (Change from baseline) | -9.4 (14.00)
  Fears/Shame (Baseline) | 49.5 (21.76)
  Fears/Shame (Change from baseline) | -14.1 (21.12)
  Nutrition (Baseline) | 12.5 (16.37)
  Nutrition (Change from baseline) | -6.3 (24.09)

17. Primary Outcome: Number of Participants With Breakthrough Angioedema Attacks
Description: A breakthrough attack was defined as an angioedema attack that occurs during long-term prevention therapy with CINRYZE (that is, between first study drug and last study drug dose). Number of participants with 1, 2, 3 or more angioedema attacks and who achieved initial improvement and complete resolution were also reported. Breakthrough angioedema attacks assessed by CINRYZE treatment, non-CINRYZE C1 INH treatment and untreated with C1-INH were reported. Here BAA refers to breakthrough angioedema attacks.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment. Number of participants evaluable for this outcome measure was reported.
Measure: Count of Participants; unit: Participants
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Participants
  Treated (CINRYZE) | 2
  Treated (NON-CINRYZE C1 INH) | 1
  Untreated | 6
  Treated (CINRYZE): One BAA | 1
  Treated (CINRYZE): Two BAA | 0
  Treated (CINRYZE): Three BAA | 1
  Treated (NON-CINRYZE C1 INH): One BAA | 0
  Treated (NON-CINRYZE C1 INH): Two BAA | 0
  Treated (NON-CINRYZE C1 INH): Three BAA | 1
  Untreated: One BAA | 1
  Untreated: Two BAA | 0
  Untreated: Three BAA | 5
  Treated (CINRYZE): Initial improvement | 2
  Treated (NON-CINRYZE C1 INH): Initial improvement | 1
  Untreated: Initial improvement | 6
  Treated (CINRYZE): Complete resolution | 2
  Treated (NON-CINRYZE C1 INH): Complete resolution | 1
  Untreated: Complete resolution | 6

18. Primary Outcome: Time From Attack Onset to Initial Improvement and Complete Resolution
Description: Time to initial improvement (TII) was calculated from the time of study drug administration to initial symptom improvement. Time to complete resolution was defined as the time from the onset of attack to complete resolution of all symptoms. Time to initial improvement and time to complete resolution as assessed by CINRYZE, non-CINRYZE and untreated were reported.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment. Number of participants evaluable for this outcome were reported.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Hours
  Treated (CINRYZE): TII: number analyzed (Participants) | 2
  Treated (CINRYZE): TII | 13.38 [4.250 to 22.500]
  Treated (NON-CINRYZE): TII: number analyzed (Participants) | 1
  Treated (NON-CINRYZE): TII | 6.42 [NA to NA] — 95% confidence interval lower and upper limits was not calculated due to insufficient number of participants.
  Untreated: TII: number analyzed (Participants) | 6
  Untreated: TII | 10.75 [8.750 to 118.000]
  Treated (CINRYZE): Complete resolution: number analyzed (Participants) | 2
  Treated (CINRYZE): Complete resolution | 40.67 [23.834 to 57.500]
  Treated (NON-CINRYZE): Complete resolution: number analyzed (Participants) | 1
  Treated (NON-CINRYZE): Complete resolution | 9.00 [NA to NA] — 95% confidence interval lower and upper limits was not calculated due to insufficient number of participants.
  Untreated: Complete resolution: number analyzed (Participants) | 6
  Untreated: Complete resolution | 61.83 [11.000 to 152.000]

19. Primary Outcome: Time From Onset of Attack to Time Treated by CINRYZE
Description: The median time from onset of attack to time treated with CINRYZE was reported.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 postbaseline efficacy assessment.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Hours | 11.97 [3.050 to 20.884]

20. Primary Outcome: Time From Treatment With CINRYZE to Initial Improvement
Description: Time to initial improvement was calculated from the time of study drug administration to initial symptom improvement. Median time from treatment with CINRYZE to initial improvement was reported.
Time Frame: Baseline up to Week 12
Population: FAS included all participants who had at least 1 post-baseline efficacy assessment.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | CINRYZE 1000 U
Number analyzed (Participants) | 8
Hours | 1.41 [1.200 to 1.617]

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 12
Arm/Group | CINRYZE 1000 U
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CINRYZE 1000 U (N=8)
Hereditary angioedema (Congenital, familial and genetic disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CINRYZE 1000 U (N=8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (3)
Seasonal allergy (Immune system disorders) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 3 (4)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Somnolence (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)
Breast disorder (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT02865720/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT02865720/SAP_001.pdf